CLINICAL TRIAL: NCT03852524
Title: Double-Blind, Randomized Trial of Peri-operative Subcutaneous Methylnaltrexone Versus Placebo for Postoperative Ileus Prevention After Adult Spinal Arthrodesis
Brief Title: Subcutaneous Methylnaltrexone Versus Placebo for Postoperative Ileus Prevention
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, H Francis Farhadi, MD, PhD, Assistant Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2018H0260
Record Dates: First submitted 2019-02-04; First posted 2019-02-25 (Actual); Results first posted 2021-10-06 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Postoperative Ileus
Keywords: Spinal Arthrodesis; Ileus; Postoperative Ileus; Adult Spinal Deformity
MeSH Terms: conditions — Ileus | interventions — methylnaltrexone

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1:1 fashion to receive methylnaltrexone or placebo. Participants will remain in the group they are randomized to for the duration of the study.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Study Arm (Experimental): The study arm will receive subcutaneous methylnaltrexone (0.15mg/kg rounded to 8 or 12 mg) before surgery and then daily, for the following three days after surgery (four doses).
  Interventions: Drug: Methylnaltrexone
- Placebo Arm (Placebo Comparator): The placebo arm will receive subcutaneous placebo before surgery and then daily, for the following three days after surgery (four doses).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Methylnaltrexone — Randomization of methylnaltrexone to placebo will be at a 1:1 ratio. Those receiving methylnaltrexone (study drug) will receive a subcutaneous dose pre-surgery and daily for three days following surgery.
  Arms: Study Arm
Other: Placebo — Randomization of methylnaltrexone to placebo will be at a 1:1 ratio. Those receiving placebo will receive a subcutaneous dose pre-surgery and daily for three days following surgery.
  Arms: Placebo Arm

SUMMARY:
This randomized controlled trial will prospectively evaluate the clinical benefit for subcutaneous methylnaltrexone (MNTX) in counteracting the obstipatory (causing constipation) effects of spinal surgery without increasing narcotic usage or otherwise disrupting the recovery course of patients. Using a double-blind randomized design, either subcutaneous MNTX (0.15 mg/kg rounded to 8 mg or 12 mg) or placebo will be administered starting before surgery and then daily for three days. Information will be collected from medical records in IHIS up to 30 days prior to surgery and then for up to 30 days after surgery.

DETAILED DESCRIPTION:
Postoperative Ileus refers to the transient interruption of propulsive motor activity of the gastrointestinal (GI) tract that prevents effective movement of its contents and tolerance of oral intake. Although POI is generally considered to significantly increase hospital stays and inpatient costs after spinal surgery, the incidence, associated risk factors, and effective preventative strategies remain poorly characterized. The proposed etiologies underlying POI are broad and remain incompletely characterized. They include post surgical sympathetic nervous system activation, inflammatory factors, and the effects of analgesics on GI tract motility. Treatment often consists of aggressive bowel regimens, nasogastric tube insertion for decompression, and the application of various laxatives, suppositories, and enemas. The widespread use of these measures is unfortunately not supported by high level evidence. The incidence of POI after spinal fusion is reported to range between 0.6 to 16.7%. This estimated range likely represents a gross underestimate of POI given the retrospective nature of studies undertaken to date. Fineberg and colleagues reported that the risk increases nearly 3-fold following anterior lumbar spinal fusions as compared to posterior surgeries. Furthermore, the only risk factors they identified to be correlated with POI is male gender, = 3 fusion levels, alcohol abuse, anemia, electrolyte abnormalities, and weight loss. Kiely and colleagues found that ileus was associated with the administration of certain intravenous solutions such as lactated ringers and sodium chloride. Interestingly, they found that albumin administration was associated with a reduced incidence of ileus postoperatively. Lee and colleagues evaluated POI following orthopedic surgery and reported an incidence of 2.1%. They found that patients who developed POI were more likely to be older, had higher blood loss during surgery, and also had higher rates of preoperative constipation. This study, however, included all types of orthopedic surgeries (not limited to spinal fusion). Early clinical studies evaluated the effectiveness of MNTX in treating opioid-induced constipation (OIC). Several clinical trials confirmed that MNTX was well tolerated and counteracted the GI effects of opioids, thereby enhancing gut motility without inhibiting their analgesic properties. Only two studies to date have evaluated the potential effectiveness of MNTX in reducing the incidence of POI following GI surgery. Both studies were unfortunately hampered by serious design flaws. Most importantly, neither study included pre-operative administration of MNTX. As such, MNTX remains at this time approved only for chronic OIC based on two double-blind, randomized, placebo-controlled trials conducted in patients with advanced illness wherein MNTX rapidly induced laxation as compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Subject is scheduled to undergo a 1 - 3 level lumbar spinal fusion for degenerative spinal conditions including neurogenic claudication and/or lumbar radiculopathy with stenosis and/or spondylolisthesis.
* Subject must be over the age of 18 years old.
* Subject has been unresponsive to conservative care for a minimum of 6 months.
* The subject must in the investigator's opinion, be psychosocially, mentally, and physically able to fully comply with this protocol and have the ability to understand and give written informed consent.

Exclusion Criteria:

* Previous Treatment with MNTX
* History of mechanical gastrointestinal obstruction
* History of OIC refractory to outpatient medical management
* Presence of a peritoneal catheter for intraperitoneal chemotherapy or dialysis
* Clinically relevant active diverticular disease
* Recent history of bowel surgery within previous 12 months
* Use of vinca alkaloids within previous four months
* Renal failure defined as Estimated Glomerular Filtration Rate (eGFR) <30 ml/min per 1.73 m^2 or requires dialysis
* Known or suspected allergy to MNTX or similar compounds (e.g. naltrexone or naloxone)
* Participation in a study with investigational products within 30 days before first dose of MNTX
* Pregnant or nursing
* Clinically important abnormalities that may interfere with participation or compliance to the study, as determined by investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2019-02-21 (Actual); Primary Completion 2021-04-04 (Actual); Study Completion 2021-05-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gifford CS, McGahan BG, Miracle SD, Minnema AJ, Murphy CV, Vazquez DE, Weaver TE, Farhadi HF. Design and feasibility of a double-blind, randomized trial of peri-operative methylnaltrexone for postoperative ileus prevention after adult spinal arthrodesis. Contemp Clin Trials. 2022 Jan;112:106623. doi: 10.1016/j.cct.2021.106623. Epub 2021 Nov 17. PMID 34798295

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Arm: Methylnaltrexone: The study arm will receive subcutaneous methylnaltrexone (0.15mg/kg rounded to 8 or 12 mg) before surgery and then daily, for the following three days after surgery (four doses).
  Methylnaltrexone: Randomization of methylnaltrexone to placebo will be at a 1:1 ratio. Those receiving methylnaltrexone (study drug) will receive a subcutaneous dose pre-surgery and daily for three days following surgery.
Period: Overall Study
Arm/Group | Study Arm: Methylnaltrexone | Placebo Arm
Started | 41 | 41
Completed | 41 | 41
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Study Arm: Methylnaltrexone | Placebo Arm | Total
Number analyzed (Participants) | 41 | 41 | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 28 | 57
  >=65 years | 12 | 13 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (10.2) | 60.8 (10.0) | 61.3 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 23 | 44
  Male | 20 | 18 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 40 | 38 | 78
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 7 | 9
  White | 38 | 34 | 72
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 41 | 41 | 82

OUTCOME MEASURES:

1. Primary Outcome: Time to First Bowel Movement
Description: The time it takes for the participant to have a bowel movement from the end of surgery.
Time Frame: 30 days post-operative
Measure: Median (Full Range); unit: hours
Arm/Group | Study Arm: Methylnaltrexone | Placebo Arm
Number analyzed (Participants) | 41 | 41
hours | 61.8 [35.7 to 93.6] | 50.7 [17.8 to 110.8]
Statistical Analysis 1: Comparison: Study Arm: Methylnaltrexone vs Placebo Arm; The sample size (41 patients per study group; 82 patients total) for this superiority trial was calculated with a power of 90% (alpha = 0.05) and based on the assumption that 50% of subjects in the placebo group would experience a bowel movement by postoperative day 3, as compared to 85% in the treatment group. Additionally, a 10% lost-to-follow up rate was assumed; Test type: Superiority; p = 0.81, Log Rank; Median Difference (Net) = 11

2. Secondary Outcome: Time to Discharge
Description: The number of hours it takes for the participant to meet all discharge criteria and be released from the hospital.(Time-to-discharge/discharge eligibility)
Time Frame: 30 Days post-operative
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Study Arm: Methylnaltrexone | Placebo Arm
Number analyzed (Participants) | 41 | 41
Hours | 105.0 [84.6 to 110.2] | 90.7 [85.4 to 111.3]

3. Secondary Outcome: Time to Discharge
Description: The time it takes for the participant to discharge
Time Frame: 30 Days post-operative
Measure: Mean (Full Range); unit: Days
Arm/Group | Study Arm: Methylnaltrexone | Placebo Arm
Number analyzed (Participants) | 41 | 41
Days | 4.29 [3.38 to 8.39] | 4.19 [3.23 to 7.69]

4. Other Pre Specified Outcome: Daily Narcotics
Description: The amount of daily narcotics (in morphine milli-equivalents) given to a patient (average of post op day 1 - 3)
Time Frame: 30 days post-operative
Measure: Median (Inter-Quartile Range); unit: MME
Arm/Group | Study Arm: Methylnaltrexone | Placebo Arm
Number analyzed (Participants) | 41 | 41
MME | 136.8 [107.9 to 168.6] | 148.5 [94.8 to 203.7]

ADVERSE EVENTS:
Time Frame: Immediately pre-operative to 30 Days post-operative
Arm/Group | Study Arm: Methylnaltrexone | Placebo Arm
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/41
Serious Adverse Events (participants affected / at risk) | 6/41 | 7/41
Other Adverse Events (participants affected / at risk) | 11/41 | 7/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Arm: Methylnaltrexone (N=41) | Placebo Arm (N=41)
Disorientation/ Hallucinations secondary to alcohol withdrawal (Psychiatric disorders) | 0 (0) | 1 (1)
Migratory artheralgias/ gout flare up (Immune system disorders) | 0 (0) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Wound Dehiscence (Infections and infestations) | 0 (0) | 1 (1)
Stroke (Vascular disorders) | 0 (0) | 1 (1)
Non-ST-elevation myocardial infarction (NSTEMI) (Cardiac disorders) | 0 (0) | 1 (1)
Altered mental status (AMS) (Psychiatric disorders) | 1 (1) | 1 (1)
hypoxemia, loss of response (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Syncope; dehydration; Fracture- Right foot (Social circumstances) | 1 (1) | 0 (0) — Fall out of bed
Post-Operative Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) — Subject refused SOC bowel regimen
urinary tract infection (UTI) and hyponatremia (Renal and urinary disorders) | 1 (1) | 0 (0)
Atrial fibrillation (also called AFib or AF) with rapid ventricular rate or response (RVR).; (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Arm: Methylnaltrexone (N=41) | Placebo Arm (N=41)
> 3 bowel movements in 1 day (Gastrointestinal disorders) | 4 (4) | 1 (1)
AMS and emesis during attempted bowel movement. (Psychiatric disorders) | 1 (1) | 0 (0)
Wound dehiscence / drainage from incision (Infections and infestations) | 2 (2) | 2 (2)
Hemoglobin drop (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Intraoperatively, a Cerebrospinal Fluid (CSF) leak was noted. (Surgical and medical procedures) | 1 (1) | 0 (0)
Diagnosis of Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Post-operative illeus (Gastrointestinal disorders) | 1 (1) | 1 (1)
increasing pain with concern for infection without drainage or dis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hypotension, syncope (Cardiac disorders) | 0 (0) | 1 (1)
Kidney Disease Improving Global Outcomes Stage III (kidney disease) (Renal and urinary disorders) | 0 (0) | 1 (1)
left airspace disease concerning for brewing aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-20): https://cdn.clinicaltrials.gov/large-docs/24/NCT03852524/Prot_SAP_000.pdf
  • Informed Consent Form (2020-11-20): https://cdn.clinicaltrials.gov/large-docs/24/NCT03852524/ICF_001.pdf